CLINICAL TRIAL: NCT02780284
Title: Gut Microbiota, Butyrate, Inflammation and Physical Activity: A Pilot Study Among Individuals at High Risk for Colorectal Cancer
Brief Title: Microbiome, Exercise Tracking Study: Among Individuals at High Risk for Colorectal Cancer
Acronym: METS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAP1611
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: Gut Microbiota; Butyrate; Physical activity
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention (Experimental): Subjects at higher risk of developing colorectal cancer will maintain the current level of activity during the first 4 weeks and exercise 150 minutes per week during the last 4 weeks. During the entire study, subjects will wear a Fitbit device on their wrist.
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — 150 minutes per week of moderate intensity cardiovascular exercise. The exercise sessions will include a minimum of 30 minutes of exercise each day, 3 to 5 times per week for a total of 150 minutes of exercise per week.

SUMMARY:
The purpose of this study has 2 aims:

Aim 1: To demonstrate the feasibility of recruiting and retaining adults at high risk of colorectal cancer to a physical activity intervention trial. Investigators hypothesize that it will be possible to recruit and retain this patient population to a physical activity intervention trial.

Aim 2: To demonstrate the feasibility of collecting, processing, storing stool samples and analyzing the gut microbiome data. Investigators hypothesize that all of these steps are feasible.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer-related deaths in the U.S. and is the third most common cancer in men and women. CRC risk factors include genetic predisposition, host factors and modifiable lifestyle behaviors (e.g., diet, physical activity, obesity). There are very limited data on the differences in the gut microbiota among populations at different levels of CRC risk, as well as the effects of behavioral interventions to alter the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English or Spanish;
2. At high risk of developing colorectal cancer;
3. No history of colorectal cancer, including germ-line heritable colorectal cancers such as Familial Adenomatous Polyposis (FAP) and Hereditary Nonpolyposis Colorectal Cancer (HNPCC);
4. No use of antibiotics in the previous 3 months; or current regular use of antibiotics
5. Access to either smart phone or computer; and
6. Currently physically inactive.

Exclusion Criteria:

Any criterion not met under inclusion.

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants retained at the end of study | 8 weeks
  To demonstrate the feasibility of recruiting and retaining adults at high risk of colorectal cancer to a physical activity intervention trial

SECONDARY OUTCOMES:
Percentage of participants with collected, processed, and analyzed stool samples | 8 weeks
  To demonstrate the feasibility of collecting, processing, storing stool samples and analyzing gut microbiome data

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, ND, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided